CLINICAL TRIAL: NCT04242355
Title: Effects of Repetitive Transcranial Magnetic Stimulation on Neural and Behavioral Facets of Social Cognition in Autism Spectrum Disorder
Brief Title: Transcranial Magnetic Stimulation on Neural and Behavioral Facets of Social Cognition in Autism Spectrum Disorder
Acronym: TMSinASD
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Yale University (Other)
Responsible Party: Principal Investigator, James C. McPartland, Associate Professor of Child Psychiatry and Psychology, Yale University
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 2000021846
Record Dates: First submitted 2020-01-15; First posted 2020-01-27 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2025-08

CONDITIONS: Autism Spectrum Disorder
Keywords: TMS
MeSH Terms: conditions — Autism Spectrum Disorder | interventions — Transcranial Magnetic Stimulation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Transcranial Magnetic Stimulation - real (Active Comparator): Participants will receive active TMS during their study visit
  Interventions: Behavioral: Transcranial Magnetic Stimulation (TMS)
- Transcranial Magnetic Stimulation - sham (Placebo Comparator): Participants will receive sham stimulation during their study visit simulating TMS
  Interventions: Behavioral: Transcranial Magnetic Stimulation (TMS)

INTERVENTIONS:
Behavioral: Transcranial Magnetic Stimulation (TMS) — Subjects will receive both active and sham TMS in a randomized crossover assignment involving two study sessions

SUMMARY:
This study will evaluate the effects of repetitive Transcranial Magnetic Stimulation (rTMS) on neural and behavioral facets of social cognition in Autism Spectrum Disorder (ASD). Participant visits will include a baseline assessment of neuropsychological, cognitive and behavioral function, and an EEG (electroencephalogram) and eye-tracking session to measure neural and visual attentional social response before and after administration of TMS.

DETAILED DESCRIPTION:
Broad ranging social cognition difficulties are hallmark areas of impairment in autism spectrum disorder (ASD), and they are subserved by specific neural systems underpinning social perception and processing that are recognized to be atypical in ASD. Considering the neurodevelopmental nature of the disorder, and the recent findings regarding aberrant neuroplasticity in ASD, repetitive transcranial magnetic stimulation (rTMS) holds promise to directly modulate brain activity in these systems. The objective of this research proposal is to utilize a multimodal approach to provide a proof-of-concept for the ability of rTMS to (a) influence functioning in the brain systems involved in social ASD symptomatology and (b) modify associated social cognitive behaviors in adults with ASD. Toward achieving this objective, we propose to assess critical aspects of social cognition using the electroencephalogram (EEG), event-related potentials (ERPS), eye-tracking (ET), and behavioral tasks prior to and following a single rTMS session to provide preliminary insight into the potential of rTMS as a tool to modify social brain function in cognitively able adults with ASD.

ELIGIBILITY:
Inclusion Criteria:

* individuals between the ages of 18 and 40 years old with typical development or with a diagnosis of autism spectrum disorder.
* able to participate in an EEG and eye-tracking experiment

Exclusion Criteria:

* Participants reporting significant head trauma or serious brain illness
* Participants with major psychiatric illness that would preclude completion of study measures.
* Participants with a history of serious medical illness, stroke, seizures, epileptiform EEG abnormalities, or family history of seizures.
* Participants taking prescription medications that may affect cognitive processes under study.
* Participants who have taken alcohol or recreational drugs within the preceding 24 hours.
* Females of known/suspected pregnancy or who test positive on a pregnancy test.
* Participants with a history of metalworking or injury by shrapnel or metallic objects are also exclude

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 100 (Estimated)
Dates: Start 2019-07-01 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2027-07 (Estimated)

PRIMARY OUTCOMES:
right lateralized N170 latency to upright faces | Measures will be recorded for the duration of their visit, an expected average of 4-5 hrs.
  EEG brain response to faces as measured by the N170 component in milliseconds

SECONDARY OUTCOMES:
proportion of visual attention to the eye region of the face | Measures will be recorded for the duration of their visit, an expected average of 4-5 hrs.
  visual attention to the eye region of the face as measured by eye tracking in seconds
The Benton Face Recognition Task | Measures will be recorded for the duration of their visit, an expected average of 4-5hrs
  The total Benton score will be used to assess the ability to recognize and discriminate among faces

CONTACTS AND LOCATIONS:
Locations (1):
- Yale University, New Haven, Connecticut, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Rossi S, Hallett M, Rossini PM, Pascual-Leone A; Safety of TMS Consensus Group. Safety, ethical considerations, and application guidelines for the use of transcranial magnetic stimulation in clinical practice and research. Clin Neurophysiol. 2009 Dec;120(12):2008-2039. doi: 10.1016/j.clinph.2009.08.016. Epub 2009 Oct 14. PMID 19833552
- [Background] Huang YZ, Edwards MJ, Rounis E, Bhatia KP, Rothwell JC. Theta burst stimulation of the human motor cortex. Neuron. 2005 Jan 20;45(2):201-6. doi: 10.1016/j.neuron.2004.12.033. PMID 15664172
- [Background] Allison T, Puce A, McCarthy G. Social perception from visual cues: role of the STS region. Trends Cogn Sci. 2000 Jul;4(7):267-278. doi: 10.1016/s1364-6613(00)01501-1. PMID 10859571
- [Background] McPartland J, Dawson G, Webb SJ, Panagiotides H, Carver LJ. Event-related brain potentials reveal anomalies in temporal processing of faces in autism spectrum disorder. J Child Psychol Psychiatry. 2004 Oct;45(7):1235-45. doi: 10.1111/j.1469-7610.2004.00318.x. PMID 15335344
- [Background] Dawson G, Toth K, Abbott R, Osterling J, Munson J, Estes A, Liaw J. Early social attention impairments in autism: social orienting, joint attention, and attention to distress. Dev Psychol. 2004 Mar;40(2):271-83. doi: 10.1037/0012-1649.40.2.271. PMID 14979766
- [Background] Oberman LM, Rotenberg A, Pascual-Leone A. Use of transcranial magnetic stimulation in autism spectrum disorders. J Autism Dev Disord. 2015 Feb;45(2):524-36. doi: 10.1007/s10803-013-1960-2. PMID 24127165
- [Background] Abujadi C, Croarkin PE, Bellini BB, Brentani H, Marcolin MA. Intermittent theta-burst transcranial magnetic stimulation for autism spectrum disorder: an open-label pilot study. Braz J Psychiatry. 2018 Jul-Sep;40(3):309-311. doi: 10.1590/1516-4446-2017-2279. Epub 2017 Dec 11. PMID 29236921
- [Background] Ni HC, Hung J, Wu CT, Wu YY, Chang CJ, Chen RS, Huang YZ. The Impact of Single Session Intermittent Theta-Burst Stimulation over the Dorsolateral Prefrontal Cortex and Posterior Superior Temporal Sulcus on Adults with Autism Spectrum Disorder. Front Neurosci. 2017 May 9;11:255. doi: 10.3389/fnins.2017.00255. eCollection 2017. PMID 28536500